CLINICAL TRIAL: NCT06124014
Title: Cranial Electrotherapy Stimulation (CES) for the Treatment of Generalized Anxiety Disorder (GAD) in Young Adults: Double-Blind Sham-Controlled Randomized Clinical Trial
Brief Title: CES for the Treatment of GAD in Young Adults
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Electromedical Products International, Inc. (Industry)
Collaborators: University of North Carolina, Chapel Hill (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 22-3341
Record Dates: First submitted 2023-10-20; First posted 2023-11-09 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-02

CONDITIONS: Generalized Anxiety Disorder
Keywords: CES
MeSH Terms: conditions — Generalized Anxiety Disorder

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Cranial Electrotherapy Stimulation (CES) (Experimental): Alpha-Stim AID ® is an FDA-cleared device for the treatment of anxiety that delivers CES through two earclip electrodes.
  Interventions: Device: At-Home Stimulation
- Sham Cranial Electrotherapy Stimulation (CES) (Sham Comparator): The device for sham stimulation is physically identical and delivers a non-therapeutic dose of stimulation to replicate salient features of device usage.
  Interventions: Device: At-Home Stimulation

INTERVENTIONS:
Device: At-Home Stimulation — The stimulation paradigm in this trial consists of six weeks of daily, 60-minute at-home stimulation sessions.

SUMMARY:
The purpose of this research study is to study cranial electrotherapy stimulation (CES) to determine its effects on symptoms of anxiety in people with generalized anxiety disorder (GAD) between the ages of 18 - 21 years of age.

DETAILED DESCRIPTION:
This study examines (1) the efficacy of CES with the Alpha-Stim AID ® for the treatment of GAD in young adults (18-21 years of age) in a double-blind, sham-controlled parallel group single-site clinical trial of 130 participants.

Participants will be randomized into receiving either active CES (at least 200uA, up to 500uA at 0.5Hz, 60 minutes daily for six weeks) or sham CES with the Alpha-Stim AID ® device at-home. Clinical assessments of anxiety symptoms are performed at Screening (for eligibility), Baseline, Follow-Up 1 (at completion of intervention, 6 weeks after initial stimulation), and Follow-Up 2 (12 weeks after initial stimulation). Additional assessments of depression symptoms and quality of life are included. Resting-state EEG will be collected at baseline and Follow-Up 1 (in up to 60 participants) for exploratory investigation of mechanism of action.

ELIGIBILITY:
Inclusion Criteria:

* Capable of signing informed consent form.
* Stated willingness to comply with all study procedures and availability for the duration of the study including refraining from changes to treatment unless medically indicated and communicated to the study team.
* Aged 18 - 21 at time of screening visit.
* Diagnosis of generalized anxiety disorder (GAD).
* At least mild-to-moderate symptom severity, as indicated by scores of 15 or higher on the clinician-administered HAM-A at the screening visit.
* Concurrent psychiatric medications are allowed. Participants will be required to maintain a sable dose of medications, or remain medication free, for 2 weeks prior to the screening visit, except for antidepressants for which the period of stable dose is 4 weeks prior to screening visit. Concurrent psychotherapy is allowed.
* People of reproductive potential must be willing to use effective contraception (evidence-based hormonal or barrier methods) for at least 1 month prior to the screening visit and agree to use such a method during study participation.

Exclusion Criteria:

Time-frames are determined relative to the screening visit.

* Current (any) or previous (> 7 stimulation sessions in last 6 weeks) use of a CES device.
* Inability to tolerate the required minimum stimulation amplitude (200 uA) during the initial device training at the baseline visit.
* Experimental or clinical brain stimulation such as deep brain stimulation or transcranial magnetic stimulation for any indication (current or within 60 days prior to screening visit).
* Implanted medical device that uses electricity anywhere in the body.
* Diagnosis (based on MINI) of bipolar I or II (past or current), moderate or severe alcohol use disorder (within 12 months prior to screening visit), moderate or severe (non-alcohol) substance use disorder (within 12 months prior to screening visit), psychotic disorder (current or lifetime), major depressive disorder with psychotic features, bipolar I with psychotic features, anorexia nervosa.
* Epilepsy (current or history). History of febrile childhood seizures and non-epileptic seizures are allowed.
* Pregnant or breast-feeding.
* Enrollment in clinical trial for any condition (current or within 60 days prior to screening visit).
* Hospitalization for any reason (current or past 2 weeks).
* Self-harming behaviors (current or within two years prior to screening visit).
* Higher than low suicide risk on the Columbia Suicide Severity Rating Scale (C-SSRS).
* Known cardiac abnormality or clinically significant heart disease.
* Anything that would make participation in the study unsafe or medically unadvisable in the assessment of a study clinician.

Ages: 18 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 130 (Estimated)
Dates: Start 2024-01-26 (Actual); Primary Completion 2025-12-17 (Actual); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Hamilton Anxiety Rating Scale (HAM-A) change | 42 days
  Change in HAM-A between six-week follow-up (FU1) and baseline (D1); minimum value is 0, maximum value is 56. Higher scores indicate worse outcome.

SECONDARY OUTCOMES:
Hamilton Anxiety Rating Scale (HAM-A) change | 84 days
  Change in HAM-A between twelve-week follow-up (FU2) and D1; minimum value is 0, maximum value is 56. Higher scores indicate worse outcome.
Beck Anxiety Inventory (BAI) Change | 42 days
  Change in BAI between FU1 and D1; minimum value is 0, maximum value is 63. Higher scores indicate worse outcome.
Beck Anxiety Inventory (BAI) Change | 84 days
  Change in BAI between FU2 and D1; minimum value is 0, maximum value is 63. Higher scores indicate worse outcome.
Generalized-Anxiety Disorder 7-item (GAD-7) Change | 42 days
  Change in GAD-7 between FU1 and D1; minimum value is 0, maximum value is 21. Higher scores indicate worse outcome.
Generalized-Anxiety Disorder 7-item (GAD-7) Change | 84 days
  Change in GAD-7 between FU2 and baseline D1; minimum value is 0, maximum value is 21. Higher scores indicate worse outcome.
Response/Remission of anxiety | 42 days
  Response/remission rates based on HAM-A scores from FU1 versus baseline D1
Response/Remission of anxiety | 84 days
  Response/remission rates based on HAM-A scores from FU2 versus baseline D1
Change in Clinical Global Impression Scale (CGI) | 42 days
  Change in CGI from FU1 to D1; CGI scale contains two scoring components, 1) Severity of Illness (0-7) and 2) Global Improvement (0-7). Higher scores in component 1 indicate worse symptoms while higher numbers in component 2 indicate worse clinical outcomes.
Change in Clinical Global Impression Scale (CGI) | 84 days
  Change in CGI from FU2 to baseline D1; CGI scale contains two scoring components, 1) Severity of Illness (0-7) and 2) Global Improvement (0-7). Higher scores in component 1 indicate worse symptoms while higher numbers in component 2 indicate worse clinical outcomes.
Change in Quality of Life Enjoyment and Satisfaction Questionnaire, short form (Q-LES-Q-SF) | 42 days
  Change in Q-LES-Q-SF from FU1 to D1; minimum value is 14, maximum value is 70. Higher scores indicate better outcome.
Change in Quality of Life Enjoyment and Satisfaction Questionnaire, short form (Q-LES-Q-SF) | 84 days
  Change in Q-LES-Q-SF from FU2 to D1; minimum value is 14, maximum value is 70. Higher scores indicate better outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Samantha Meltzer-Brody, MD, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- Carolina Center for Neurostimulation, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Barclay TH, Barclay RD. A clinical trial of cranial electrotherapy stimulation for anxiety and comorbid depression. J Affect Disord. 2014 Aug;164:171-7. doi: 10.1016/j.jad.2014.04.029. Epub 2014 Apr 21. PMID 24856571
- [Background] Bandelow B, Michaelis S. Epidemiology of anxiety disorders in the 21st century. Dialogues Clin Neurosci. 2015 Sep;17(3):327-35. doi: 10.31887/DCNS.2015.17.3/bbandelow. PMID 26487813
- [Background] Goodwin RD, Weinberger AH, Kim JH, Wu M, Galea S. Trends in anxiety among adults in the United States, 2008-2018: Rapid increases among young adults. J Psychiatr Res. 2020 Nov;130:441-446. doi: 10.1016/j.jpsychires.2020.08.014. Epub 2020 Aug 21. PMID 32905958
- [Background] Hajek A, Sabat I, Neumann-Bohme S, Schreyogg J, Barros PP, Stargardt T, Konig HH. Prevalence and determinants of probable depression and anxiety during the COVID-19 pandemic in seven countries: Longitudinal evidence from the European COvid Survey (ECOS). J Affect Disord. 2022 Feb 15;299:517-524. doi: 10.1016/j.jad.2021.12.029. Epub 2021 Dec 15. PMID 34920039
- [Background] Garakani A, Murrough JW, Freire RC, Thom RP, Larkin K, Buono FD, Iosifescu DV. Pharmacotherapy of Anxiety Disorders: Current and Emerging Treatment Options. Front Psychiatry. 2020 Dec 23;11:595584. doi: 10.3389/fpsyt.2020.595584. eCollection 2020. PMID 33424664
- See also: Link to more information and study recruitment for interested potential participants. — https://www.carolinaneurostimulation.org/open-studies.html